CLINICAL TRIAL: NCT04359316
Title: Efficacy and Safety of Azithromycin Compared to the Base Therapeutic Regiment of Hydroxychloroquine in Moderate to Severe COVID-19: A Randomized, Controlled, Double-Blind, Clinical Trial
Brief Title: Azithromycin in Hospitalized COVID-19 Patients
Acronym: AIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyed Sina Naghibi Irvani, MD, MPH, MBA, Senior Researcher., Dr., Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Azithromycin in COVID-19
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Novel Coronavirus; Hydroxychloroquine; Chloroquine; Azithromycin
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Intervention Model Description: The present study is a randomized, double-blind, placebo-controlled, clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Shahid Modarres Medical Education Center and Hospital in Tehran. Patients will be randomly assigned to the two arms of the study and after completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin (Experimental)
  Interventions: Drug: Hydroxychloroquine; Drug: Azithromycin
- Hydroxychloroquine (Active Comparator)
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — This Drug will be used in all arms as mandated by our governmental guidelines.
Drug: Azithromycin — This will be drug only used in the intervention arm of our study, designed mainly to assess the additional efficacy and safety of Azithromycin in COVID-19 patients.
  Arms: Azithromycin

SUMMARY:
The present study is a randomized, double-blind, controlled, clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Shahid Modarres Medical Education Center and Hospital in Tehran. Patients will be randomly assigned to the two arms of the study and after completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.

DETAILED DESCRIPTION:
Chloroquine has been a broadly-utilized anti-malaria agent which back in 2006, had been proved to be a powerful wide-spectrum antiviral. Moreover, Chloroquine has the characteristics of anti-inflammatory and immune-modulatory by inhibiting the production of TNF-α along with IL-6. In the first half of February, a study illustrated puissant inhibition of SARS-CoV-2 by Chloroquine, when taking two 500-mg tablets of it by mouth per day; similar to some clinical studies in China through this outbreak. According to the news briefing of a study, it was indicated that chloroquine phosphate actually outdo the control treatment in inhibition of pneumonia exacerbation, improving lung imaging findings, and curtailing the disease course. Another study evaluated the possible doses of CQ and HCQ to find the optimized dose in treatment of COVID-19. They revealed that while within in-vitro settings Hydroxychloroquine is more potent than chloroquine. As a conclusion, they suggested a 800 mg daily dose of hydroxychloroquine, followed by an overall maintenance dose of 400 mg per day divided in two separate doses, which was three-fold more potent compared to the 500 mg twice daily administration of chloroquine in 5 days. The new study published in 16th March, pointed out that hydroxychloroquine was notably effectual in eradicating SARS-CoV-2 from the nasopharynx. Currently the evidence is quite inconclusive about the effectiveness or comparative effectiveness of either HCQ or CQ. Moreover, CQ has recently become scarce and even unavailable for ordering due to a huge demand for it, all because of a significant interest gained as a potential medicinal alternative for the management of COVID-19. In spite of all, the primary experience in China and France is propitious for the potential role of chloroquine, or alternatively hydroxychloroquine, for managing COVID-19.

The reported clinical benefits of the combination of hydroxychloroquine and azithromycin for patients with COVID-19 come either from media reports or nonrandomized trials with small numbers of participants (<100 patients). The documented benefit of hydroxychloroquine with or without azithromycin is very limited, especially in severe disease. While these medications, individually or in combination, may prove efficacious, these benefits need to be established with randomized clinical trials prior to widespread adoption of these treatments.

The present study is a randomized, double-blind, controlled, clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Shahid Modarres Medical Education Center and Hospital in Tehran. Patients will be randomly assigned to the two arms of the study and after completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* COVID-19 Confirmed Cases (Either RT-PCR or CT Scan Confirmed).
* Tympanic Temperature of ≥37.5 AND at least one of the following: Cough, Sputum production, nasal discharge, myalgia, headache or fatigue) on admission.
* Time of onset of the symptoms should be acute ( Days ≤ 10).
* SpO2 ≤ 93%
* Respiratory Rate ≥ 22

Exclusion Criteria:

* Refusal to participate expressed by patient or legally authorized representative if they are present.
* Patients with prolonged QT or PR intervals, Second or Third Degree heart block and Arrhythmias.
* Patients using drugs with potential interaction with Azithromycin or Hydroxychloroquine.
* Pregnant or lactating women.
* History of alcohol or drug addiction in the past 5 years.
* Blood ALT/AST levels > 5 times the upper limit of normal on laboratory results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-05-03 (Estimated); Study Completion 2020-05-05 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | From date of randomization until 14 days later.
  Improvement of two points on a seven-category ordinal scale (recommended by the World Health Organization: Coronavirus disease (COVID-2019) R&D. Geneva: World Health Organization) or discharge from the hospital, whichever came first.

SECONDARY OUTCOMES:
Mortality | From date of randomization until 14 days later.
  If the patient dies, we have reached an outcome.
SpO2 Improvement | Days 1, 2, 3, 4, 5, 6, 7 and 14.
  Pulse-oxymetry
Incidence of new mechanical ventilation use | From date of randomization until 14 days later.
  Incidence of new mechanical ventilation use (Rate)
Duration of hospitalization | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 14 days.
  Duration of hospitalization (Days)
Cumulative incidence of serious adverse events | Days 1, 2, 3, 4, 5, 6, 7 and 14.
  With incidence of any serious adverse effects, the outcome has happened.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Fathi, MD, Study Chair — Shahid Beheshti University of Medical Sciences; Sasan Tavana, MD, Study Director — Shahid Beheshti University of Medical Sciences; Nasser Malekpour Alamdari, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Mehran Lack, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Nader Markazi, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Sanaz Zargar Balaye Jam, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Seyed Sina Naghibi Irvani, MD, MPH, MBA, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shahid Modarres Hospital, Shahid Beheshti University of Medical Sciences and Health Services, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided
There is no further information.